CLINICAL TRIAL: NCT00370981
Title: A Four-arm, Randomized, Double-blind, Parallel, Placebo-controlled Exploratory Study of Pagoclone 0.15mg, 0.30mg, and 0.60mg in Men With Primary Premature Ejaculation.
Brief Title: Exploratory Study of Pagoclone in Men With Premature Ejaculation.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IP456-040
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2007-02

CONDITIONS: Premature Ejaculation
Keywords: investigational drug; ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — pagoclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.15 mg (Experimental)
  Interventions: Drug: pagoclone
- 0.30 mg (Experimental)
  Interventions: Drug: pagoclone
- 0.60 mg (Experimental)
  Interventions: Drug: pagoclone
- PBO (Placebo Comparator)
  Interventions: Drug: pagoclone

INTERVENTIONS:
Drug: pagoclone

SUMMARY:
The purpose of this study is to evaluate pagoclone in the treatment of premature ejaculation.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effect of 3 dose levels of pagoclone (0.15 mg, 0.30 mg, and 0.60 mg) versus placebo on intravaginal ejaculation latency time (IELT) male patients with primary premature ejaculation.

ELIGIBILITY:
Inclusion Criteria:

* A male regularly experiencing premature ejaculation
* 18 to 55 yrs old
* In a Stable relationship with one woman for at least 6 months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100
Dates: Start 2006-07; Primary Completion 2006-07 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Intravaginal ejaculation latency time (IELT)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Urology Centers of Alabama, PC, Homewood, Alabama
  - SD Uro-Research, San Diego, California
  - Urology Research Options, Aurora, Colorado
  - Urology Associates, PC, Denver, Colorado
  - Connecticut Clinical Research Center, Waterbury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - Davis Clinic, PC, Indianapolis, Indiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - AccuMed Research Associates, Garden City, New York
  - Urological Surgeons of Long Island, PC, Garden City, New York
  - Center for Urologic Research of WNY, Williamsville, New York
  - Metrolina Urology Clinic, Charlotte, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Johnny B. Roy, MD Private Practice, Edmond, Oklahoma
  - Mobley Research Center, Houston, Texas